CLINICAL TRIAL: NCT04387097
Title: Postoperative Drip-infusion of Remifentanil for Preventing Remifentanil-induced Hyperalgesia- a Retrospective Observative Study
Brief Title: Drip-infusion of Remifentanil for RIH
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yi-hsuan Huang, Principal Investigator, Tri-Service General Hospital
Other Study IDs: TSGHIRB No: 2-108-05-135
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hyperalgesia
Keywords: Remifentanil; Hyperalgesia; Drip-infusion
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil; Infusions, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gradual withdrawal following by drip-infusion of remifentanil: In the end of the surgery, gradual withdrawal of remifentanil was prescribed until the endotracheal tube was extubated. Following by drip-infusion of remifentanil for 30 minutes was administered immediately after tracheal extubation.
  Interventions: Drug: remifentanil
- gradual withdrawal of remifentanil: In the end of the surgery, gradual withdrawal of remifentanil was prescribed until the endotracheal tube was extubated.

INTERVENTIONS:
Drug: remifentanil — postoperative drip-infusion of remifentanil
  Other Names: drip-infusion
  Groups: gradual withdrawal following by drip-infusion of remifentanil

SUMMARY:
The development of remifentanil-induced hyperalgesia (RIH) is an unpleasant experience for surgical patients. An alternative management, gradual withdrawal of remifentanil was effective in prevention of RIH. The investigators designed a simple modality to assess if under withdrawal of remifentanil and further drip-infusion of remifentanil immediately after extubation affected postoperative pain score, the requirement of rescue analgesics, and adverse effects.

DETAILED DESCRIPTION:
In clinical practice, the gradual withdrawal of remifentanil during surgery is unsatisfied. Thus, the investigators conducted a simple modality in a single center retrospective cohort study to assess how under baseline gradual withdrawal of remifentanil and further drip infusion of remifentanil immediately after extubation affected postoperative pain score and use of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score of I-III patients receiving total intravenous anesthesia

Exclusion Criteria:

* The use of inhalation agents or propofol combined with inhalation anesthesia
* Pregnancy
* Previous substance abuse
* Known allergies to opioids, propofol or any drugs used in the study
* History of neuropsychiatric disorder
* Age < 20 years or > 80 years

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving surgery with age between 20-80 years
Sampling Method: Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
comparison of the numeric rating scale (NRS) between 2 groups | one hour
  NRS scores is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.
requirement for rescue analgesics | one hour
  postoperative requirement for rescue analgesics

SECONDARY OUTCOMES:
type of surgery | three hours
  type of surgery in both groups
surgical site | three hours
  surgical site in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Yi-hsuan Huang, MD, Principal Investigator — Tri-Service General Hospital and National Defense Medical Center
Locations (1):
- TriService General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Comelon M, Raeder J, Stubhaug A, Nielsen CS, Draegni T, Lenz H. Gradual withdrawal of remifentanil infusion may prevent opioid-induced hyperalgesia. Br J Anaesth. 2016 Apr;116(4):524-30. doi: 10.1093/bja/aev547. Epub 2016 Mar 1. PMID 26934941
- [Result] Saxena S, Gonsette K, Terram W, Huybrechts I, Nahrwold DA, Cappello M, Barvais L, Engelman E. Gradual withdrawal of remifentanil delays initial post-operative analgesic demand after thyroid surgery; double-blinded, randomized controlled trial. BMC Anesthesiol. 2019 Apr 25;19(1):60. doi: 10.1186/s12871-019-0731-9. PMID 31027480